CLINICAL TRIAL: NCT03137459
Title: STAMP: Sharing and Talking About My Preferences
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1604017648; 1R01NR016007-01 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Advanced Care Planning (ACP)
Keywords: Transtheoretical Model (TTM)
MeSH Terms: interventions — Transtheoretical Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TTM (Experimental): Participants enrolled at the intervention site will receive four contacts, at baseline, two, four and six months. Each of the first three contacts consists of an integrated assessment and intervention feedback report, using an expert system.
  Interventions: Behavioral: Transtheoretical Model (TTM) of health behavior change
- Usual Care (Active Comparator): Participants enrolled in control sites will receive four assessment contacts on the same schedule and in the same manner as the participants enrolled in intervention sites.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Transtheoretical Model (TTM) of health behavior change — Participants are assessed for four different behaviors that together represent complete ACP engagement: communication with loved ones about views on quality of life versus quantity of life, communication with clinicians about views on quality of life versus quantity of life, assignment of a health care surrogate, and completion of a living will. The system takes the results of the assessment and results in an individualized feedback report. For individuals in early stages of change for a given behavior, the feedback focuses on changing attitudes, a necessary prerequisite for changing behavior, by addressing common barriers and by reminding individuals they can engage in small steps.
  Arms: TTM
Other: Usual Care — Participants are assessed for four different behaviors that together represent complete ACP engagement: communication with loved ones about views on quality of life versus quantity of life, communication with clinicians about views on quality of life versus quantity of life, assignment of a health care surrogate, and completion of a living will. Participants in this group will not receive any components of the TTM intervention.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to examine the effect of an individually transtheoretical model (TTM) tailored intervention on the completion of advance care planning (ACP) behaviors.

DETAILED DESCRIPTION:
This will be a randomized controlled trial examining the effect of an individually TTM-tailored intervention on the proportion of middle-age and older persons recruited from primary care practices who complete four ACP behaviors (completion of a living will, assignment of a health care proxy, and communication with loved ones and with their clinician about views on quality versus quantity of life) over six months, compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be community-dwelling persons with an upcoming primary care visit in the study's practice settings.

Exclusion Criteria:

* Severe hearing impairment, defined as being unable to participate in a telephone conversation.
* Severe visual impairment, defined as being unable to read large-print materials.
* Moderate to severe cognitive impairment, defined as either a diagnosis of dementia and/or short-term recall of <2/3 objects at 2 minutes.
* Primary language other than English.
* Having completed all of the four ACP behaviors that are the focus of this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Fried, MD, Principal Investigator — Internal Medicine: Geriatrics: Claude D. Pepper Older Americans Independence Center; Dorothy Adler Geriatric Assessment Center
Locations (1):
- Northeast Medical Groups, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fried TR, Paiva AL, Redding CA, Iannone L, O'Leary JR, Zenoni M, Risi MM, Mejnartowicz S, Rossi JS. Effect of the STAMP (Sharing and Talking About My Preferences) Intervention on Completing Multiple Advance Care Planning Activities in Ambulatory Care : A Cluster Randomized Controlled Trial. Ann Intern Med. 2021 Nov;174(11):1519-1527. doi: 10.7326/M21-1007. Epub 2021 Aug 31. PMID 34461035
- [Derived] Fried TR, Redding CA, Martino S, Paiva A, Iannone L, Zenoni M, Blakley LA, Rossi JS, O'Leary J. Increasing engagement in advance care planning using a behaviour change model: study protocol for the STAMP randomised controlled trials. BMJ Open. 2018 Aug 10;8(8):e025340. doi: 10.1136/bmjopen-2018-025340. PMID 30099405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 ambulatory internal medicine practices, matched in pairs according to practice type and percentage of patients age 65+, non-White, and receiving Medicaid
Pre-assignment Details: Because randomization occurred at the level of the practice, participants' assignment to group was determined before any information was known about them. However, there were participants who were excluded from they study before beginning any study procedures. These included: 1 matched set of practices was excluded for failing to meet minimum enrollment with 12 participants; 6 participants consented in error; 25 participants refused the baseline interview.
Groups:
- STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report: Participants enrolled at the intervention site will receive four contacts, at baseline, two, four and six months. Each of the first three contacts consists of an integrated assessment and intervention feedback report, using an expert system.
  Transtheoretical Model (TTM) of health behavior change: Participants are assessed for four different behaviors that together represent complete advance care planning (ACP) engagement: communication with loved ones about views on quality of life versus quantity of life, communication with clinicians about views on quality of life versus quantity of life, assignment of a health care surrogate, and completion of a living will. The system takes the results of the assessment and results in an individualized feedback report. For individuals in early stages of change for a given behavior, the feedback focuses on changing attitudes, a necessary prerequisite for changing behavior, by addressing common barriers and by reminding individuals they can engage in small steps.
Period: 2-month Assessment
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Started | 455 | 454
Completed | 387 | 412
Not Completed | 68 | 42
Not completed — Withdrawal by Subject | 13 | 3
Not completed — Unable to reach | 42 | 32
Not completed — Refused assessment | 7 | 5
Not completed — Acutely ill | 6 | 2
Period: 4-month Assessment
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Started | 442 | 451
Completed | 364 | 405
Not Completed | 78 | 46
Not completed — Death | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Unable to reach | 44 | 29
Not completed — Refused assessment | 24 | 10
Not completed — Acutely ill | 2 | 3
Period: 6-months
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Started | 434 | 447
Completed | 413 | 430
Not Completed | 21 | 17
Not completed — Lost to Follow-up | 14 | 11
Not completed — Death | 0 | 2
Not completed — Refused assessment | 6 | 3
Not completed — Acutely ill | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report: Participants enrolled at the intervention site will receive four contacts, at baseline, two, four and six months. Each of the first three contacts consists of an integrated assessment and intervention feedback report, using an expert system.
  Transtheoretical Model (TTM) of health behavior change: Participants are assessed for four different behaviors that together represent complete ACP engagement: communication with loved ones about views on quality of life versus quantity of life, communication with clinicians about views on quality of life versus quantity of life, assignment of a health care surrogate, and completion of a living will. The system takes the results of the assessment and results in an individualized feedback report. For individuals in early stages of change for a given behavior, the feedback focuses on changing attitudes, a necessary prerequisite for changing behavior, by addressing common barriers and by reminding individuals they can engage in small steps.
- Total: Total of all reporting groups
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care | Total
Number analyzed (Participants) | 455 | 454 | 909
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.5) | 67.8 (8.0) | 68.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 262 | 554
  Male | 163 | 192 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 441 | 439 | 880
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 76 | 91 | 167
  White | 352 | 339 | 691
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 9 | 10 | 19
Education [Count of Participants; unit: Participants]
  <=12th grade | 137 | 96 | 233
  >12th grade | 318 | 358 | 676
Employment [Count of Participants; unit: Participants]
  Employed | 157 | 194 | 351
  Unemployed | 298 | 260 | 558
Baseline stage of change: living will [Count of Participants; unit: Participants]
  Precontemplation | 64 | 86 | 150
  Contemplation | 224 | 224 | 448
  Preparation | 59 | 21 | 80
  Action/maintenance | 108 | 120 | 228
  Missing | 0 | 3 | 3
Baseline stage of change: healthcare agent [Count of Participants; unit: Participants]
  Precontemplation | 69 | 99 | 168
  Contemplation | 227 | 217 | 444
  Preparation | 76 | 31 | 107
  Action/maintenance | 83 | 105 | 188
  Missing | 0 | 2 | 2
Baseline stage of change: communication about quality versus quantity of life [Count of Participants; unit: Participants]
  Precontemplation | 80 | 112 | 192
  Contemplation | 60 | 46 | 106
  Preparation | 11 | 5 | 16
  Action/maintenance | 304 | 289 | 593
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Four ACP Activities: Communication With Loved Ones About Quality Versus Quantity of Life, Completion of a Living Will, Assignment of a Healthcare Agent, and Confirmation of Documents in the Electronic Health Record.
Description: The primary outcome of the study is to assess the proportion of participants that have completed the four ACP behaviors. The measure will be coded as a binary outcome where 'yes' indicates the completion of all 4 behaviors and 'no' indicates no completing the 4 behaviors.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Number analyzed (Participants) | 455 | 454
Participants | 64 | 37
Statistical Analysis 1: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Risk Difference (RD) = .059, 95% CI 2-sided [.014 to .105] — Analysis performed using GEE to account for clustering of participants within practices
Statistical Analysis 2: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.14 to 2.93] — Determined using mixed effects models, accounting for clustering of participants in practices and adjusting for unbalanced covariates: education, employment, stage of change for each ACP behavior

2. Secondary Outcome: Number of Participants Who Complete a Living Will
Time Frame: 6-months
Population: Participants who had not completed a living will at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Number analyzed (Participants) | 347 | 334
Participants | 99 | 68
Statistical Analysis 1: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Risk Difference (RD) = .082, 95% CI 2-sided [.014 to .150] — Adjusted for clustering
Statistical Analysis 2: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.39, 95% CI 2-sided [.96 to 2.0] — Accounting for clustering and adjusted for covariates as described in primary outcome

3. Secondary Outcome: Number of Participants Who Assign a Healthcare Agent
Time Frame: 6 months
Population: Individuals who had not assigned a healthcare agent at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Number analyzed (Participants) | 372 | 349
Participants | 122 | 68
Statistical Analysis 1: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Risk Difference (RD) = .133, 95% CI 2-sided [.066 to .201] — Accounting for clustering
Statistical Analysis 2: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.22 to 2.47] — Accounting for clustering and adjusted for covariates as presenting for primary outcome

4. Secondary Outcome: Number of Participants Who Communicate With a Loved One About Quality Versus Quantity of Life
Time Frame: 6 months
Population: Individuals who had not communicated about quality versus quantity of life at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
Number analyzed (Participants) | 151 | 165
Participants | 93 | 90
Statistical Analysis 1: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Risk Difference (RD) = .070, 95% CI 2-sided [-.05 to .188]
Statistical Analysis 2: Comparison: STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.15, 95% CI 2-sided [.72 to 1.85] — Accounting for clustering and adjusting for covariates as described for primary outcome

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | STAMP: Computer-Tailored Intervention Consisting of Assessment With Feedback Report | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/455 | 0/454
Serious Adverse Events (participants affected / at risk) | 0/455 | 0/454
Other Adverse Events (participants affected / at risk) | 0/455 | 0/454

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03137459/Prot_SAP_000.pdf